CLINICAL TRIAL: NCT02651103
Title: Changes in Cerebral Oxygenation Based on Intraoperative Ventilation Strategy
Status: Completed | Type: Observational
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chairman: Professor of Anesthesiology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB15-01073
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Results first posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2017-12

CONDITIONS: Posterior Spinal Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Posterior spinal fusion: Patients undergoing spinal fusion surgery
  Interventions: Device: NIRS

INTERVENTIONS:
Device: NIRS — Cerebral oxygenation monitor which is standard of care for this surgery.

SUMMARY:
The proposed research aims to investigate how different ventilation strategies may affect cerebral tissue oxygenation in the pediatric population. It will contribute to the literature exploring the NIRS monitoring device which is becoming increasingly utilized in a variety of anesthetic and critical care settings. It may help to guide clinical practice regarding optimal ventilation strategies, and how ventilation may be altered to correct suboptimal cerebral tissue oxygenation.

This prospective study will include 50 patients undergoing posterior spinal fusion that requires placement of an arterial cannulation. There will be no change in the anesthetic or perioperative care of these patients. Tissue and cerebral oxygenation will be monitored using near infrared spectroscopy (NIRS).

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing spinal surgery

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing posterior spinal fusion
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Tobias, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Posterior Spinal Fusion
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Posterior Spinal Fusion
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Cerebral Oxygenation Values Throughout the Procedure
Description: Measured on the NIRS cerebral oxygenation monitor attached to the patient
Time Frame: prior to induction of anesthesia in the awake patient and following four ventilation strategies (average time frame of 15 mins. to 5 hours)
Measure: Mean (Standard Deviation); unit: rSO2
Arm/Group | Posterior Spinal Fusion
Number analyzed (Participants) | 30
rSO2
  Phase 1 | 83 (8)
  Phase 2 | 79 (8)
  Phase 3 | 81 (9)
  Phase 4 | 83 (8)

ADVERSE EVENTS:
Time Frame: through study completion, an average of 2 years
Description: All-Cause Mortality, Serious, or Other (non-serious) Adverse Events were monitored/assessed, but none observed
Arm/Group | Posterior Spinal Fusion
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT02651103/Prot_SAP_000.pdf